CLINICAL TRIAL: NCT00220857
Title: Rapid Protection of the Gastroduodenal Mucosa Against Aspirin-Induced Damage by Rabeprazole
Brief Title: Rabeprazole Protection of Aspirin Induced Gastric Damage.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TU4504
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Normal Subjects
Keywords: Rabeprazole; Nonsteroidal Antiinflammatory Drugs; Gastric erosions
MeSH Terms: interventions — Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole

SUMMARY:
To determine the effectiveness of rabeprazole in preventing or decreasing acute gastroduodenal injury caused by therapeutic doses of aspirin in a placebo-controlled, randomized, double-blind parallel group study.

DETAILED DESCRIPTION:
Thirty (30) eligible normal subjects will be randomized to one of two study groups: rabeprazole 20 mg OD (n=15) or placebo OD (n=15). Both rabeprazole and identically appearing placebo will be given to Temple from Janssen Pharmaceuticals. The randomization schedule will be prepared by John Gaughan, PhD of Temple University School of Medicine Department of Biostatistics using a random number generator. The coded medications will be dispensed by Temple's Department of Pharmacy. Study subjects and the investigators will be blinded as to the subject receiving either placebo or rabeprazole. The sealed code will not be broken until after the data analysis.

Study subjects will be admitted to the Temple Clinical Research Center for the duration of the study. Appendix I has the study time line. Study subjects will arrive at the CRC at 6:00 A.M. on study day 1. Female subjects will have a urine pregnancy test performed. Blood tests will be obtained for salicylate and alcohol levels. Each study subject will receive a single dose of study drug (rabeprazole or placebo) at 7:00 A.M. on study days 1, 2 and 3-one hour before breakfast on days 1 and 3 and 90 minutes before breakfast on study day 2. All research subjects will receive aspirin (ASA), 325 mg tablets as 2 tablets with 8 oz. water every 4 hours at 8:30 A.M., 12:30 P.M., 4:30 P.M., 8:30 P.M., 12:30 A.M. and 4:30 A.M. daily for study days 1, 2 and 3 (a total of 3900 mg aspirin per day). Esophagogastroduodenoscopy will be performed at 8:00 A.M. on the mornings of days 2 and 4; that is, 24 hours and 72 hours after initiation of aspirin and test drug. During each endoscopy, the maximum number of submucosal hemorrhages and erosions in an endoscopic field from the anterior and posterior walls of the antrum will be counted. In addition, a Lanza score will be assigned for each endoscopic examination (Appendix II). Endoscopic photographs will be obtained for each endoscopic examination. A blood sample will be obtained at 7:00 A.M. on study days 2, 3 and 4 for measurement of hemoglobin and serum salicylate. Meals will be standardized as follows for each day of the study:

Breakfast: 8:00 A.M. (study days 1 and 3); 8:30 A.M. (study day 2) 2 eggs, 2 slices of soft white bread, 4 oz unsweetened orange juice Lunch: 1:00 P.M. (study days 1, 2 and 3) Turkey sandwich, 2 slices of wheat bread, lettuce, tomato, 1 orange, 8 oz apple juice Dinner: 6:00 P.M. (study days 1, 2 and 3) Two plain hamburgers, ketchup, mustard, lettuce and tomato; tossed green salad with thousand island dressing, 1 cup of French fries, 8 oz whole milk Snack: 10:00 P.M. (study days 1, 2 and 3) 4 graham crackers, 4 oz orange juice

If the Lanza score reaches 4 for any subject indicating widespread involvement of the stomach with submucosal hemorrhages, erosions, or ulcerations, that subject will not receive any more aspirin, but continue with study drug of placebo or rabeprazole. If this was detected on day 2 of the study, the subject will continue to receive the study drug with the repeat study endoscopy on day 4. If the Lanza score day 4 (the end of the study) is 4, the subject will be treated with rabeprazole 20 mg po qd for one month. If there was an ulcer, a repeat upper endoscopy will then be performed at 4 weeks to ensure healing.

ELIGIBILITY:
Thirty (30) normal subjects will be recruited.

Inclusion criteria:

* A normal subject must be between 18 and 60 years of age with no history of gastrointestinal disease, gastroduodenal surgery, upper gastrointestinal symptoms or cardiopulmonary disease of any kind.

Exclusion Criteria:

* Normal subjects should have not ingested a salicylate, nonsteroidal antiinflammatory drug, histamine-2 receptor antagonist, proton pump inhibitor, misoprostol or carafate within one month of entering this study.
* He/she should not have participated in an investigational study within 3 months of this protocol.
* Pregnant women and women not using an accepted method of birth control will be excluded.
* Patients will be excluded who are allergic to aspirin and NSAIDs, who have an intolerance to aspirin and NSAIDs, who have a history of asthma and/or nasal polyps.
* Patients will be excluded if they have a history of gastric ulcers, duodenal ulcers, gastrointestinal bleeding, or bleeding disorder, clotting disorder.
* Patients will be excluded who actively abuse alcohol, as defined by greater than three twelve ounce beers or greater than three drinks containing hard liquor per day.
* Patients with a history of intracranial bleeding and/or brain trauma will be excluded from this research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Gastric mucosal abnormalities

SECONDARY OUTCOMES:
Hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fisher, MD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Medicine, Philadelphia, Pennsylvania, United States